CLINICAL TRIAL: NCT05034341
Title: Does Prehabilitation Improve Outcomes in Patients Undergoing Complex Spine Fusion Surgery?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution and unable to complete study.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202000987; OCR39834 (Other: UF OnCore)
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Lumbar Spine Injury; Spinal Fusion; Frailty; Prehabilitation; Nutritional Supplementation; Functional Outcome
Keywords: Frailty; Prehabilitation; Perioperative Outcomes
MeSH Terms: conditions — Spinal Injuries; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Prehabilitation Arm (Experimental): The Multimodal Prehabilitation group will receive:
  * An exercise program focusing on aerobic exercise as well as strength training. Sessions will be supervised by a physical therapist, 2 times a week for a minimum of 6-8 weeks in addition to a home exercise program. Patients' compliance will be monitored by phone each week.
  * Protein supplements in the form of protein shakes at a dose of 1.2-1.5 gram per kg daily for 6-8 weeks. Protein supplements will be calculated based on ideal body weight and will be given to the patient with instructions on specific use. Diabetic patients will receive protein supplements that are sugar-free.
  * Pain and Neuroscience Education: Per University of Florida Health Pain and Neuroscience program at Shands hospital.
  * Standard Clinical Care: Preoperative medical optimization and management, referral to medical specialties as deemed necessary with a focus on preoperative cognitive assessment.
  Interventions: Other: Multimodal Prehabilitation
- Standard Clinical Care Comparison Arm (Active Comparator): The Standard Clinical Care Comparison group will receive:
  * Education related to preoperative activity and home based exercise program.
  * Standard preoperative consultation with anesthesiology: Preoperative medical optimization and management, referral to medical specialties as deemed necessary with focus on preoperative cognitive assessment.
  * A final preoperative visit before surgery where a second set of functional assessment will be implemented
  Interventions: Other: Standard Pre-Surgical Clinical Care

INTERVENTIONS:
Other: Multimodal Prehabilitation — In addition to Standard Clinical Care
  Behavioral - An exercise program focusing on aerobic exercise as well as strength training. Sessions will be supervised by a physical therapist, 2 times a week for a minimum of 6-8 weeks in addition to home exercise program. They will also participate in a single session of Cognitive-Behavioral Therapy and will receive an educational pamphlet about Pain and Neuroscience Education.
  Dietary Supplement - Protein supplements in the form of protein shakes at a dose of 1.2-1.5 gram per kg daily for 6-8 weeks. Protein supplements will be calculated based on ideal body weight and will be given to the patient with instructions on specific use. Diabetic patients will receive protein supplements that are sugar free.
  Arms: Multimodal Prehabilitation Arm
Other: Standard Pre-Surgical Clinical Care — * Education related to preoperative activity and home-based exercise program.
  * Standard preoperative consultation with anesthesiology: Preoperative medical optimization and management, referral to medical specialties as deemed necessary with focus on preoperative cognitive assessment.
  Arms: Standard Clinical Care Comparison Arm

SUMMARY:
A novel prehabilitation method has been implemented at our institution to decrease perioperative outcome complications for frail complex spine fusion surgery patients. The goal of this randomized trial is to evaluate whether this prehabilitation program improves preoperative functional status of frail spine disease patients and benefits patients in their postsurgical outcomes.

DETAILED DESCRIPTION:
Background:

Patients with degenerative lumbar spine disease who are candidates for spine surgery may experience multiple adverse effects from the prolonged conservative and non-operative management of chronic low back pain. Due to the aging population, there is an increased demand for lumbar spine surgery in the geriatric population. At the time these patients are candidates for surgery, they might encounter the results of the conservative management including disabling pain, catastrophizing, and Kinesiophobia. The chronicity of the spine condition and the associated pain may result in functional disability, poor nutrition, and poor pain management, all of which may result in a multisystemic impact on their overall health in the form of frailty. Prehabilitation has been studied in the past to evaluate its impact on the postoperative outcomes for patients scheduled for abdominal surgery, cardiac surgery, and thoracic surgery. Currently, there are a few trials evaluating the impact of prehabilitation in spine surgery. However, there are limited data on the impact of prehabilitation on frail geriatric patients undergoing spine surgery and whether prehabilitation will impact frail patients' preoperative and postoperative functional recovery and pain management.

Based on the current literature, the investigator will hypothesize that prehabilitation will improve frail geriatric patients' preoperative and postoperative functional capacity as assessed by a six-minute walk test and will minimize the incidence of postoperative complications. In addition, the investigator will also hypothesize that prehabilitation in the form of a multimodal approach (physical exercise, nutritional, pain, and neuroscience education) will increase the chances of discharge to home in the postoperative setting, and as a result will lead to a decrease overall healthcare expenditure and total costs.

Specific Aims:

1. Does Multimodal Prehabilitation improve frail patients' preoperative functional capacity before spine surgery?
2. Does Multimodal Prehabilitation improve frail patients' postoperative outcomes after spine surgery?
3. Does Multimodal Prehabilitation improve frail patients' postoperative functional capacity after spine surgery?

The investigator will hypothesize that Multimodal Prehabilitation (physical, nutritional, and cognitive) improves frailty, functional capacity, and perioperative outcomes after spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Frailty score of 3 or more (based on Johns Hopkins Frailty Assessment).
* Age 55 and older
* Elective Lumbar or thoracolumbar Spine Fusion Surgery

Exclusion Criteria:

* Emergency surgery
* Time-sensitive surgery
* Spine trauma, tumor, or infection
* Physical condition that limits exercise: Lower extremity amputation, hemiplegia or hemiparesis, stroke with residual weakness, symptomatic severe cardiac disease (for example: severe aortic stenosis, unstable angina)
* Patient refusal
* Severe cognitive dysfunction preventing participation or consenting.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Frailty Assessment | Baseline up to 3 months
  Johns Hopkins Frailty Assessment
6 Minute Walk Test | Baseline up to 3 months
  Distance and Percent Predicted Distance Travelled by Walking for 6 Minutes and then evaluating their performance in comparison to normal population. Also, measuring the the symptoms of fatigue and severity of dyspnea on exertion

CONTACTS AND LOCATIONS:
Overall Officials: Basma Mohamed, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Health of University of Florida, Gainesville, Florida, United States